CLINICAL TRIAL: NCT02238561
Title: The Cost in Oxygen of Surgical Trauma (CO2ST) - a Feasibility Study of the Non-invasive Measurement of Oxygen Delivery and Consumption After Major Abdominal Surgery
Brief Title: The Cost in Oxygen of Surgical Trauma
Status: Completed | Type: Observational
Sponsor: University Hospital Plymouth NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 14/P/123
Record Dates: First submitted 2014-09-09; First posted 2014-09-12 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-02

CONDITIONS: Oxygen Consumption (V̇O2); Oxygen Delivery (DO2); Post-operative Complications
Keywords: non-invasive; measurement of oxygen; consumption; delivery; post-operative complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Elective major abdominal surgery: Patients undergoing elective major open or laparoscopic abdominal surgery at Plymouth Hospitals National Health Service (NHS) Trust (PHNT)

SUMMARY:
The investigators will examine the relationship between post-operative oxygen consumption (using non-invasive measurement technology ) and complications in patients having contemporary major abdominal surgery. The investigators hypothesis is that major surgery may trigger a physiological stress response that results in an increase in post-operative metabolic demand and oxygen consumption (V̇O2) which must be met by an increased oxygen delivery (DO2).

1. To determine the feasibility of non-invasive measurement of oxygen consumption (V̇O2) using indirect calorimetry in a cohort of patients
2. To determine the feasibility of non-invasive measurement of oxygen delivery (DO2) in the same cohort using non-invasive measures of cardiac output, oxygen saturation and haemoglobin (pulse wave transit time and co-oximetry techniques)

DETAILED DESCRIPTION:
Prospective observational study of non-invasive measurements of V̇O2 and DO2 pre-operatively and at 8 time points in the 48 hours postoperatively in a cohort of 40 patients undergoing elective major abdominal surgery (both open and laparoscopic) with a pre-operative cardiopulmonary exercise testing (CPET).

As pilot work examining the relationship between post-operative oxygen consumption and complications in patients having contemporary major abdominal surgery , the investigators need to define and grade the severity of complications. The Post-Operative Morbidity Survey (POMS) is a simple outcome scale designed to record the incidence of clinically important complications - specifically complications likely to keep a patient in hospital. A POMS score performed on Day 5 is likely to be discriminative between patients who are recovering well, and those who are developing complications. POMS is easily performed, has good internal validity and is predictive of a prolonged length of stay. POMS is not a simple additive scale; however patients with POMS score of 1 or greater are highly likely to remain in hospital, whereas those with a score of 0 are likely to be able to go home.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged 18 or over.
* Undergoing elective major open or laparoscopic abdominal surgery.

Exclusion Criteria:

* Refusal to participate
* Requirement for post-operative ventilation
* Requirement of inspired oxygen concentrations (FiO2) > 28% to maintain oxygen saturations ≥ 90%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective major open or laparoscopic abdominal surgery at Plymouth Hospitals NHS Trust (PHNT)
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
postoperative morbidity score (POMS) | Day 5 post surgery
  The Post-Operative Morbidity Survey (POMS) is a simple outcome scale designed to record the incidence of clinically important complications - specifically complications likely to keep a patient in hospital. A POMS score performed on Day 5 is likely to be discriminative between patients who are recovering well, and those who are developing complications. POMS is easily performed, has good internal validity and is predictive of a prolonged length of stay. POMS is not a simple additive scale; however patients with POMS score of 1 or greater are highly likely to remain in hospital, whereas those with a score of 0 are likely to be able to go home.

SECONDARY OUTCOMES:
Length of hospital stay | estimated average length of hospital stay of 5 - 7 days
  The number of days the patient is in hospital following surgery
Unplanned admission to critical care. | Participants will be followed for the duration of hospital stay, an expected average of 5 - 7 days
  We are looking at admission to critical care that was not arranged pre-operatively - a certain proportion of patients are routinely admitted to critical care because of medical co-morbidities. We are looking for those patients who were deemed fit enough not to need critical care post-operatively who subsequently need admission there, and the length of their stay there.
Returns to the operating theatre | Number of events during Hospital admission (estimated average length of hospital stay of 5 - 7 days)
  The number of times a patient has to be returned to the operating theatre during their index admission.
Hospital readmission | Within 30 days of discharge from hospital
  Number of readmissions to hospital following discharge elated to the patients surgery
Mortality | Up to 30 days following hospital discharge
  Patient mortality rate following surgery up to 30 days following discharge

CONTACTS AND LOCATIONS:
Overall Officials: Adam Kimble, BSc(Hons), MSc, MBBS, MRCS, Principal Investigator — University Hospital Plymouth NHS Trust
Locations (1):
- Plymouth Hospitals NHS Trust, Plymouth, Devon, United Kingdom